CLINICAL TRIAL: NCT00105612
Title: Improving Informed Consent in Alzheimer's Disease Research
Brief Title: Memory Aid for Informed Consent in Alzheimer's Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized
Other Study IDs: IA0070; 1R01AG020627-01A2 (NIH)
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease; Aging
Keywords: Informed Consent; Memory Aid
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Device: Memory and Organizational Aid
Behavioral: Standard Informed Consent Process — The informed consent protocol for a hypothetical early-phase drug trial will be administered by a trained interviewer in the patient's home

SUMMARY:
The purpose of this trial is to test whether a memory and organizational aid in the form of a document that summarizes and simplifies a study's key points can improve the decision-making abilities and competency of mild to early moderate Alzheimer's disease (AD) patients.

DETAILED DESCRIPTION:
Studies of mild to moderate Alzheimer's disease (AD) patients reveal substantial variation in their ability to participate in an informed consent process. No published data show techniques that help an AD patient to participate in an informed consent. This research will address this issue by performing a randomized trial to test whether a memory and organizational aid can improve the decision-making abilities and competency of AD patients.

This study will recruit 80 patients with mild to early moderate AD, and 30 non-demented elderly persons. The informed consent protocol for a hypothetical early-phase drug trial will be administered by a trained interviewer in the patient's home. The AD patients will be randomized to receive either the standard informed consent process or the intervention of the standard informed consent process plus the memory and organizational aid. All non-demented elderly individuals will receive the standard informed consent process. The interviewer will administer the protocol to participants and ask questions that will assess participant capacity to understand, appreciate, reason, and make a choice concerning enrollment in the hypothetical study.

ELIGIBILITY:
Inclusion Criteria:

* Live within one hour drive of the University of Pennsylvania's Memory Disorders Clinic
* Education equivalent to 6th grade level
* Corrected visual acuity of at least 20/70
* Speak English
* Diagnosed with possible or probable AD, or non-demented
* MMSE (Mini Mental State Exam) >= 18

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110
Dates: Start 2004-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
MacArthur Competency Assessment Tool for Clinical Research (MacCAT-CR) to quantify decision making abilities

SECONDARY OUTCOMES:
Participant competency

CONTACTS AND LOCATIONS:
Overall Officials: Jason Karlawish, MD, Principal Investigator — University of Pennsylvania Institute on Aging
Locations (1):
- University of Pennsylvania, Memory Disorders Clinic, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Marson DC, Ingram KK, Cody HA, Harrell LE. Assessing the competency of patients with Alzheimer's disease under different legal standards. A prototype instrument. Arch Neurol. 1995 Oct;52(10):949-54. doi: 10.1001/archneur.1995.00540340029010. PMID 7575221
- [Background] Kim SY, Caine ED, Currier GW, Leibovici A, Ryan JM. Assessing the competence of persons with Alzheimer's disease in providing informed consent for participation in research. Am J Psychiatry. 2001 May;158(5):712-7. doi: 10.1176/appi.ajp.158.5.712. PMID 11329391
- [Background] Sachs GA, Stocking CB, Stern R, Cox DM, Hougham G, Sachs RS. Ethical aspects of dementia research: informed consent and proxy consent. Clin Res. 1994 Oct;42(3):403-12. No abstract available. PMID 7955902
- [Background] Karlawish JH, Casarett DJ, James BD. Alzheimer's disease patients' and caregivers' capacity, competency, and reasons to enroll in an early-phase Alzheimer's disease clinical trial. J Am Geriatr Soc. 2002 Dec;50(12):2019-24. doi: 10.1046/j.1532-5415.2002.50615.x. PMID 12473015
- [Background] Appelbaum PS, Grisso T. The MacArthur Competence Assessment Tool - Clinical Research. Sarasota, FL: Professional Resources Press, 2000.
- [Derived] Rubright J, Sankar P, Casarett DJ, Gur R, Xie SX, Karlawish J. A memory and organizational aid improves Alzheimer disease research consent capacity: results of a randomized, controlled trial. Am J Geriatr Psychiatry. 2010 Dec;18(12):1124-32. doi: 10.1097/JGP.0b013e3181dd1c3b. PMID 20808101